CLINICAL TRIAL: NCT03557970
Title: A Phase 2 Open-Label Study of the CSF-1R Inhibitor JNJ-40346527 in Patients With Relapsed/Refractory Acute Myeloid Leukemia (AML)
Brief Title: JNJ-40346527 in Treating Participants With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not enough enrollment to determine efficacy
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Janssen, LP (Industry); The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Elie Traer, MD PhD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00017583; NCI-2018-00869 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00017583 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — JNJ-40346527; Pharmacogenomic Variants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (JNJ-40346527) (Experimental): Participants receive JNJ-40346527 PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Edicotinib; Other: Pharmacokinetic Study

INTERVENTIONS:
Drug: Edicotinib — Given PO
  Other Names: JNJ-40346527
Other: Pharmacokinetic Study — Correlative studies
  Other Names: PHARMACOKINETIC; PK Study

SUMMARY:
This phase II trial studies how well edicotinib (JNJ-40346527) works in treating participants with acute myeloid leukemia that has come back or does not respond to treatment. JNJ-40346527 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

Evaluate preliminary efficacy of JNJ-40346527 in participants with relapsed/refractory AML.

I. Best objective response rate (> PR).

SECONDARY OBJECTIVES:

Assess safety and survival associated with JNJ-40346527 to treat participants with relapsed/refractory AML. Assess the duration of disease response associated with JNJ-40346527.

I. Overall incidence of treatment-related and non-treatment related toxicity. II. Duration of response. III. 12-month event-free survival. IV. 12-month overall survival.

EXPLORATORY OBJECTIVES:

I. Evaluate the pharmacokinetics of JNJ-40346527 and effective inhibition of CSF-1R in marrow aspirates using plasma inhibitory assays, with established CSF-1R-sensitive cell lines.

II. Identify the effect of JNJ-40346527 on leukemia cells and the immune microenvironment.

III. Identify and quantify the specific subpopulation of cells that express CSF-1R in participants and correlate these with clinical response to JNJ-40346527.

IV. Analyze the frequency of mutations using genomic deoxyribonucleic acid (DNA) from leukemia participants to determine if there is a genetic signature that predicts response to JNJ-40346527.

V. Using ribonucleic acid (RNA) sequencing (RNAseq), identify an expression signature in CSF-1R+ cells that predicts patient response.

VI. Evaluate the effect of JNJ-40346527 on immune cell populations (cytotoxic T cells, etc.) and phospho-signaling proteins by mass cytometry (CyTOF) analysis in pre- and post-treatment samples in order to identify biomarkers that predict patient response and prioritize potential combination strategies for future clinical trials.

VII. Determine how leukemia cells change in response to CSF-1R inhibition by assessing cells collected pre- and post-treatment using an ex vivo sensitivity to a panel of small molecule inhibitors to determine what new drug sensitivities may emerge in AML cells after CSF-1R inhibition.

OUTLINE:

Participants receive JNJ-40346527 orally (PO) twice a day (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up within 2 weeks, at 4-6 weeks until death or minimum of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ability to understand and the willingness to sign a written informed consent document.
* 2. Age >= 18 years at time of informed consent. Both men and women and members of all races and ethnic groups will be included.
* 3. Morphologically documented relapsed/refractory AML as defined by World Health Organization (WHO) criteria after at least 1 prior therapy for AML with the exception of hydroxyurea, and not felt to have curative treatment options per treating physician, or the patients themselves are unwilling to consider curative treatment options.
* 4. Sufficient and viable bone marrow aspirate or peripheral blood collection to use for the ex vivo sensitivity assay.
* 5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* 6. Women must not be pregnant or breastfeeding. Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to start of study drug administration.
* 7. Participants must agree to use an adequate method contraception.
* 8. Must be able to take oral medications.
* 9. Adequate organ function as defined by the following:

  1. Serum creatinine =< 2 x the upper limit of normal (ULN), or glomerular filtration rate > 20 ml/min as calculated by Cockcroft-Gault formula.
  2. Serum potassium, magnesium, and calcium (corrected for albumin) within institutional normal limits or can be corrected with supplementation.
  3. Total serum bilirubin =< 2.5 x ULN.
  4. Serum aspartate transaminase (AST) and/or alanine transaminase (ALT) =< 2.5 x ULN.

Exclusion Criteria:

* 1. Diagnosis of acute promyelocytic leukemia (APL, or AML M3 subtype).
* 2. Active central nervous system involvement with AML.
* 3. Concurrent active malignancy with expected survival of less than 1 year. For example, candidates with treated skin cancers, prostate cancer, breast cancer, etc. without metastatic disease are candidates for therapy since their expected survival exceeds that of relapsed or refractory AML. All subjects with concurrent malignancies will be reviewed by the principal investigator (PI) prior to enrollment.
* 4. Clinically significant graft versus host disease (GVHD) or active GVHD requiring initiation or escalation of treatment within 28-day screening period.
* 5. Clinically significant coagulation abnormality, such as disseminated intravascular coagulation.
* 6. Participants who are currently receiving any other investigational agents.
* 7. Previous treatment with CSF-1R kinase inhibitor or CSF-1R blocking antibody.
* 8. Known clinically significant liver disease defined as ongoing drug-induced liver injury, chronic active hepatitis C (HCV), chronic active hepatitis B (HBV), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, portal hypertension, or history of autoimmune hepatitis.
* 9. Untreated HIV or active hepatitis C detectable by polymerase chain reaction (PCR), or chronic hepatitis B (patients positive for hepatitis B core antibody who are receiving intravenous immunoglobulin (IVIG) are eligible if hepatitis B [HepB] polymerase chain reaction [PCR] is negative).
* 10. Known history of cerebrovascular accident, myocardial infarction, or intracranial hemorrhage within 2 months of enrollment.
* 11. Clinically significant surgery within 2 weeks of enrollment.
* 12. Per PI discretion, active infection that is not well controlled by antibacterial or antiviral therapy.
* 13. Cancer-directed therapy within 2 weeks prior to starting treatment, with the exception of hydroxyurea, which is allowed to control white blood cell count. Hydroxyurea will be weaned as soon as clinically feasible.
* 14. Unwillingness to receive infusion of blood products.
* 15. Drugs that affect the CYP3A4 systems are allowed and essential for cancer patients, including anti-fungals but should be used with caution.
* 16. Patients with uncontrolled white blood cell count (defined as > 50 K/cu mm not controlled with hydrea).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elie Traer, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for this study were recruited from within the hematology and oncology practices participating research sites.
  There were 8 consented patients that were deemed screen failures and thus not enrolled on this trial. The reasons for screen failures were: patient chose alternative treatment (n=3), patient had insufficient sample for the ex vivo drug screen (n=3), patient was too sick to participate in the trial (n=1), and patient withdrew consent (n=1).
Pre-assignment Details: All enrolled participants were included in the study and assigned to 1 of 2 arms according to their ex vivo sensitivity to study drug. Consented patients with indeterminate ex vivo sensitivity were considered screen failures.
  Although this was designed as a 2-arm trial (for purposes of stopping early for futility at the end of stage 1 of the study and of correlating pre-treatment ex vivo sensitivity with post-treatment clinical response), the study drug regimen was identical in the 2 arms.
Groups:
- Assay Positive: Participants with ex vivo sensitivity to study drug according to a cell viability assay performed on participant bone marrow or peripheral blood cells. Sensitivity is defined as an IC50 that is <=20% of the median IC50.
- Assay Negative: Participants lacking ex vivo sensitivity to study drug according to a cell viability assay performed on participant bone marrow or peripheral blood cells. Lack of sensitivity is defined as an IC50 that is >20% of the median IC50.
Period: Overall Study
Arm/Group | Assay Positive | Assay Negative
Started | 1 | 2
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — Study closure | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Assay Positive | Assay Negative | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Median (Full Range); unit: years] — Age at consent
  years | 72 [72 to 72] | 60 [57 to 63] | 63 [57 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Best Objective Response Rate
Description: An objective response is defined as achievement of a PR or any type of CR (CR, CRm, CRc, CRi) during a participant's first 2 cycles of study drug. Each participant's best disease response designation (amended from the IWG criteria specified by Cheson, 2003 JCO) during the first 2 cycles will be used when computing the best objective response rate. This rate will be reported alongside an exact confidence interval for each arm separately.
Time Frame: first 2 cycles of study drug
Population: According to the protocol, only those participants who have completed at least 1 cycle of study agent and have response measurements will be evaluable for objective response. Since the only participant with a recorded disease response designation did not complete 1 cycle of study drug, there are no evaluable participants for this trial's primary outcome.
Arm/Group | Assay Positive | Assay Negative
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Incidence of Treatment-related and Non-treatment Related Adverse Events Per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Description: The overall incidence of treatment-related and non-treatment-related toxicity (including serious and non-serious AEs). See the Adverse Event module of the Results section for a tabular summary of each toxicity event and associated system organ class.
Time Frame: Start of study drug until 30 days after the last dose of study drug (while the participant remains on-study), which amounted to an average of 31 days for the 3 enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Assay Positive | Assay Negative
Number analyzed (Participants) | 1 | 2
Participants
  Treatment-related AE's (any grade) | 0 | 0
  Non-treatment-related AE's (any grade) | 1 | 2

3. Secondary Outcome: Duration of Response
Description: For participants that achieve at least a partial response (PR), the length of time between start date of this response and progression.
Time Frame: achievement of >=PR through end of study
Population: No participants achieved a response while on study so duration of response cannot be computed.
Arm/Group | Assay Positive | Assay Negative
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Event-free Survival
Description: Defined for all patients of a trial; measured from the date of entry into a study to the date of relapse from PR or CR or CRi, progression, or death from any cause; patients not known to have any of these events are censored on the date they were last examined. The Kaplan-Meier method will be used to estimate event-free survival.
Time Frame: study enrollment until last on-study disease assessment
Population: EFS cannot be calculated due to a lack of disease response information.
Arm/Group | Assay Positive | Assay Negative
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival
Description: Defined for all patients of a trial; measured from the date of entry into a study to the date of death from any cause; patients not known to have died at end of study are censored on the date they were last known to be alive. The Kaplan-Meier method will be used to estimate overall survival.
Time Frame: From study enrollment until end of participant follow-up (i.e., death or last contact), with the protocol specifying that "[p]articipants will be followed … until death"
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Assay Positive | Assay Negative
Number analyzed (Participants) | 1 | 2
months | NA [NA to NA] — There were no observed deaths in this arm (i.e., the lone participant withdrew from study to transition to hospice) so median OS could not be computed. | 6.6 [NA to NA] — This arm's sample size of 2 participants (with 1 observed death) was insufficient for calculating a confidence interval for the median OS.

ADVERSE EVENTS:
Time Frame: Per protocol "from the time subject has started study drug to completion of the study.", with post- drug exposure on-study time periods of 12, 38, and 189 days (mean of 80 days) for the 3 enrolled participants
Description: Per protocol "Toxicities will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5)."
Arm/Group | Assay Positive | Assay Negative
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/2
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assay Positive (N=1) | Assay Negative (N=2)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assay Positive (N=1) | Assay Negative (N=2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bone pain (worsening) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain in extremity (General disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT03557970/Prot_SAP_000.pdf